CLINICAL TRIAL: NCT00158717
Title: A Phase 3b, Long-Term, Observational Study of the Durability of Seroconversion in Patients With Chronic Hepatitis B Virus Infection Who Have Seroconverted While Participating in a Previous Gilead-Sponsored Study of Adefovir Dipivoxil.
Brief Title: Observational Study of the Durability of Seroconversion Chronic HBV Patients Who Seroconverted in a Previous Gilead-Sponsored Study of ADV.
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Other Study IDs: GS-00-481
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Hepatitis B
Keywords: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic | interventions — adefovir dipivoxil

INTERVENTIONS:
Drug: Hepsera

SUMMARY:
To investigate the durability of HBeAg seroconversion in patients with chronic hepatitis B virus infection (HBV) who have seroconverted while participating in a previous Gilead-sponsored study of adefovir dipivoxil.

DETAILED DESCRIPTION:
The primary objective of this study is to investigate the durability of HBeAg seroconversion in patients with chronic hepatitis B virus infection (HBV) who have seroconverted while participating in a previous Gilead-sponsored study of adefovir dipivoxil.

The secondary objective of this study is to investigate the durability of HBeAg loss in patients with chronic hepatitis B virus infection (HBV) who have experienced durable HBeAg loss while participating in a previous Gilead-sponsored study of adefovir dipivoxil.

ELIGIBILITY:
Inclusion Criteria:

* Must have met all inclusion criteria and none of the exclusion criteria and must have demonstrated HBeAg seroconversion or durable HBeAg loss as defined by the protocol in one of the following Gilead-sponsored studies: GS-96-412, GS-98-437, GS-00-461 or ongoing or future Gilead-sponsored studies identified by the Sponsor to be eligible for this study. Other patients who were enrolled in a now closed Gilead-sponsored study of ADV (GS-94-404, GS-96-412 Initial Phase or GS-96-413) and had previously demonstrated seroconversion or durable HBeAg loss during their participation will be evaluated by the clinical research organization (CRO) medical monitor for participation in this study on a case by case basis.
* Have documented negative serum HBeAg with or without positive anti-HBe present at the two study visits prior to the final visit of the previous study.
* A patient who has documented negative serum HBeAg without positive anti-HBe must also have undetectable serum HBV DNA (less than 1000 copies/mL using Roche Amplicor PCR Assay) and normalized ALT (less than ULN) confirmed during these two studies.
* All patients must be able to give written informed consent and comply with requirements of this study.

Exclusion Criteria:

* Patients who seroconvert or experience durable HBeAg loss during their participation in study GS-00-480 will not be eligible.
* Any serious or active medical or psychiatric illness that, in the opinion of the investigator would interfere with patient treatment, assessment or compliance with the protocol.
* Receiving any of the excluded medications listed in the protocol.
* Inability to comply with study requirements.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who demonstrate HBeAg seroconversion or durable HBeAg loss in one of the previous Gilead-sponsored studies listed in Section 4.2 of this protocol and meet all inclusion and none of the exclusion criteria for this study will be eligible for enrollment.
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2003-04; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Durability of HBeAg seroconversion in patients with chronic hepatitis B virus infection (HBV) who have seroconverted while participating in a previous Gilead-sponsored study of adefovir dipivoxil. | Baseline to Week 144

SECONDARY OUTCOMES:
Durability of HBeAg loss in patients with chronic hepatitis B virus infection (HBV) who have experienced durable HBeAg loss while participating in a previous Gilead-sponsored study of adefovir dipivoxil. | Baseline to Week 144

REFERENCES:
- See also: Website for Gilead — http://www.Gilead.com